CLINICAL TRIAL: NCT02502877
Title: Core Temperature Variations During Midazolam vs Propofol Sedation for Neuraxial Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital da Luz, Portugal (Other)
Responsible Party: Principal Investigator, João Pedro Gouveia, Dr., Hospital da Luz, Portugal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HDLSpot1
Record Dates: First submitted 2015-07-08; First posted 2015-07-20 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Body Temperature Changes; Anesthesia
MeSH Terms: conditions — Body Temperature Changes | interventions — Midazolam; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam Group (Other): In the "midazolam group" the investigators will administer 0,05mg/kg of midazolam, being 2/3 administered before the neuraxial block and 1/3 after.
  Interventions: Drug: Midazolam; Drug: Standard; Device: SpotOn
- Propofol group (Active Comparator): In the "propofol group" the investigators will administer 0,033mg/kg of midazolam before the neuraxial block, and immediately after installation of the block the investigators will start a propofol TCI pump (Schnider model) with an effect concentration set at 1mcg/mL. This pump will be turned off at the end of the surgery.
  Interventions: Drug: Propofol; Drug: Standard; Device: SpotOn

INTERVENTIONS:
Drug: Midazolam — The investigators will administer 0,05mg/kg of midazolam, being 2/3 administered before the neuraxial block and 1/3 after.
  Other Names: A
  Arms: Midazolam Group
Drug: Propofol — The investigators will administer 0,033mg/kg of midazolam before the neuraxial block, and immediately after installation of the block the investigators will start a propofol TCI pump (Schnider model) with an effect concentration set at 1mcg/mL. This pump will be turned off at the end of the surgery.
  Other Names: B
  Arms: Propofol group
Drug: Standard — The investigators will administer to every patient: cefazolin 2g iv bolus, ketorolac 30 mg iv bolus, pantoprazole 40 mg iv bolus, paracetamol 1g iv perfusion (initiated 30 minutes before the end of surgery).
Device: SpotOn — Central temperature will be monitored with the SpotOnTM3MTM device from entering till leaving the operating room, through a sensor placed in the patient's forehead

SUMMARY:
The present study is a pilot study aiming to compare the variation in core temperature (measured through the non-invasive device Spot-OnTM3MTM) in patients submitted to neuraxial anesthesia for orthopedic procedures, during sedation with midazolam vs propofol.

DETAILED DESCRIPTION:
In this study the investigators will select 20 patients scheduled for orthopedic surgery of the knee or foot with neuraxial anesthesia (subarachnoid or sequential blocks). Sedation for these procedures with midazolam or propofol is daily practice in the investigators' department.

So the patients will be randomized, through the envelope method, in 2 groups with 10 patients each: "midazolam group" and "propofol group".

In the "midazolam group" the investigators will administer 0,05mg/kg of midazolam, being 2/3 administered before the neuraxial block and 1/3 after.

In the "propofol group" the investigators will administer 0,033mg/kg of midazolam before the neuraxial block, and immediately after installation of the block the investigators will start a propofol target-controlled infusion (TCI) pump (Schnider model) with an effect concentration set at 1mcg/mL. This pump will be turned off at the end of the surgery.

The neuraxial block will be performed inside the operating room and preferentially in lateral decubitus. The choice of drug and dosage used for the block will be left to the anesthesiologist, to mimetize day-to-day practice. The limit dermatome of sensory block will be noted.

The investigators will administer to every patient: cefazolin 2g iv bolus, ketorolac 30 mg iv bolus, pantoprazole 40 mg iv bolus, paracetamol 1g iv perfusion (initiated 30 minutes before the end of surgery).

Central temperature will be monitored with the SpotOnTM3MTM device from entering till leaving the operating room, through a sensor placed in the patient's forehead. Room temperature will be kept at 17 degrees Celsius (ºC). Patients will be warmed with a underbody forced-air blanket (BairHuggerTM3MTM) set at 38ºC and maximal flow, initiated after performing the neuraxial block and stopped right before leaving the operating room.

Data will be analyzed with the Statistical Package for the Social Sciences (SPSS) program.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for orthopedic surgery of the foot or knee
* Indication to neuraxial anesthesia
* Surgery duration > 30 minutes

Exclusion Criteria:

* Preference for deep sedation
* Preference for no sedation
* Kidney failure
* Hepatic failure
* No signed informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Mean temperature | From entering the operating room up to cutaneous closure, an expected average of 1 to 1.5 hours
  Comparison between the mean temperature in the two groups

SECONDARY OUTCOMES:
Level of sensory block, T1-12/L1-5, assessed by a blunted needle | From 5 to 10 minutes after the performance of the neuraxial block
  Top dermatome of sensory block, evaluated with a blunt needle

CONTACTS AND LOCATIONS:
Overall Officials: João Gouveia, Dr., Principal Investigator — Hospital da Luz
Locations (1):
- Hospital da Luz, Lisbon, Lisbon District, Portugal

REFERENCES:
- [Background] Sun Z, Honar H, Sessler DI, Dalton JE, Yang D, Panjasawatwong K, Deroee AF, Salmasi V, Saager L, Kurz A. Intraoperative core temperature patterns, transfusion requirement, and hospital duration in patients warmed with forced air. Anesthesiology. 2015 Feb;122(2):276-85. doi: 10.1097/ALN.0000000000000551. PMID 25603202
- [Background] Eshraghi Y, Nasr V, Parra-Sanchez I, Van Duren A, Botham M, Santoscoy T, Sessler DI. An evaluation of a zero-heat-flux cutaneous thermometer in cardiac surgical patients. Anesth Analg. 2014 Sep;119(3):543-549. doi: 10.1213/ANE.0000000000000319. PMID 25045862
- [Background] Jeong CW, Ju J, Lee DW, Lee SH, Yoon MH. Lipid-emulsion propofol less attenuates the regulation of body temperature than micro-emulsion propofol or sevoflurane in the elderly. Yonsei Med J. 2012 Jan;53(1):198-203. doi: 10.3349/ymj.2012.53.1.198. PMID 22187253
- [Background] Iden T, Horn EP, Bein B, Bohm R, Beese J, Hocker J. Intraoperative temperature monitoring with zero heat flux technology (3M SpotOn sensor) in comparison with sublingual and nasopharyngeal temperature: An observational study. Eur J Anaesthesiol. 2015 Jun;32(6):387-91. doi: 10.1097/EJA.0000000000000232. PMID 25693138